CLINICAL TRIAL: NCT05738174
Title: Theta Burst Zur Behandlung Der Alkoholabhängigkeit
Brief Title: High-dose Accelerated Theta Burst Stimulation for the Treatment of Alcohol Addiction
Acronym: TBA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Berthold Langguth, MD, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Berthold Langguth, MD, Ph.D., Prof. Dr., University of Regensburg
Organization: University of Regensburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-3261-101
Record Dates: First submitted 2023-02-07; First posted 2023-02-21 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intermittent theta burst stimulation (iTBS) (Experimental): 1200 pulses of iTBS per session with five sessions per day applied at five days (Monday-Friday) with 120% resting motor threshold
  Interventions: Device: high-dose accelerated intermittent theta burst stimulation
- sham treatment (Sham Comparator): 1200 pulses of iTBS per session with five sessions per day applied at five days (Monday-Friday) with 120% resting motor threshold with angled coil
  Interventions: Device: sham high-dose accelerated intermittent theta burst stimulation

INTERVENTIONS:
Device: high-dose accelerated intermittent theta burst stimulation — 1200 pulses of iTBS per session with five sessions per day applied at five days (Monday-Friday) with 120% resting motor threshold
  Arms: intermittent theta burst stimulation (iTBS)
Device: sham high-dose accelerated intermittent theta burst stimulation — 1200 pulses of iTBS per session with five sessions per day applied at five days (Monday-Friday) with 120% resting motor threshold with angled coil
  Arms: sham treatment

SUMMARY:
This is a two-arm randomized placebo-controlled trial in which 72 patients with alcohol addiction are treated with high-dose accelerated intermittent theta burst stimulation (TBS).

ELIGIBILITY:
Inclusion Criteria:

* alchohol dependence according to ICD-10 (F10.2)
* desire to reduce or abstain from alcohol drinking
* male or female
* 18-65 years
* residency in Germany, German speaking
* written informed consent

Exclusion Criteria:

* contraindications for transcranial magnetic stimulation (electric devices or metal parts in the body such as pacemaker)
* relevant neurological or internistic diseases according to study investigator
* treatment with TMS in the past
* participation in other trials during treatment
* pregnancy or breatfeeding
* positive breath test for alcohol
* legal care and placement in a psychiatric hospital
* co-medication with disulfiram, acamprosate, topiramate, baclofen, naltrexone, or nalmefene
* acute psychiatric comorbidity that requires inpatient treatment or medication readjustment (<1 month)
* severe chronic psychiatric illness (schizophrenia, schizoaffective disorder, bipolar disorder)
* patients who are unable to complete study questionnaires or follow-up questionnaires (in the opinion of the investigators)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Craving visual analoge scale | one week
  alcohol craving according to visual analog scale (range: 0-100; higher values = worse outcome)

SECONDARY OUTCOMES:
Craving visual analoge scale | 13 weeks
  alcohol craving according to visual analog scale (range: 0-100; higher values = worse outcome)
relapse (number of patients with alcohol relapse) | 13 weeks
  number of patients with alcohol relapse
heavy drinking days | 13 weeks
  number of heavy drinking days (four drinks for female and five drinks for male)
abstinence confidence | 13 weeks
  abstinence confidence (Kurzfragebogen zur Abstinenzzuversicht KAZ-35; only available in German; range: 0-100%; higher values = worse outcome)
degree of dependence | 13 weeks
  degree of dependence according to DSM-5 (Diagnostic and Statistical Manual of Mental Disorders) (range: mild, moderate, severe)
Fagerström Test for Nicotine Dependence | 13 weeks
  Fagerström Test for Nicotine Dependence (range: 0-10; higher values = worse outcome)
major depression inventory | 13 weeks
  Major Depression Inventory (range: 0-50; higher values = worse outcome)
World Health Organisation quality of life bref | 13 weeks
  World Health Organisation quality of life bref (range: 4-20; lower values = worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, Principal Investigator — University Hospital of Regensburg, Department of Psychiatry and Psychotherapy at the Bezirksklinikum
Locations (1):
- Department of Psychiatry and Psychotherapy, University of Regensburg, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No